CLINICAL TRIAL: NCT06316648
Title: The Effect of Preoperative Oral Whey Intake on Blood Glucose, Fasting, Thirst, Nausea and Vomiting Levels of Patients Undergoing Elective Hip Fracture Surgery: A Randomized Controlled Study
Brief Title: Whey Intake Blood Glucose, Fasting, Thirst, Nausea and Vomiting Levels of Patients Undergoing Elective Hip Fracture Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, HÜMEYRA YÜKSEL, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 210366
Record Dates: First submitted 2024-03-10; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Elective Hip Fracture Surgery
Keywords: Whey,; Fasting; Thirsts; Nausea; Vomiting
MeSH Terms: conditions — Fasting; Nausea; Vomiting | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Multidisciplinary cooperation was performed for the effective and efficient conduct of the study. In determining the patients to administer Whey according to the study's inclusion criteria, an orthopedic and traumatological specialist's support was received, as well as that of an anesthesiologist. On the other hand, the researcher cooperated with a nutritionist in preparing and assessing the Whey content to be administered to the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): At 00:00 the night before the surgery, the researcher told the patients in the control group that they could have fruit juice/water if they wanted and waited for 10 minutes. The researcher then initiated the restriction process by informing the patients that they could no longer have food/water. Fasting, thirst, blood glucose and nausea-vomiting evaluations applied to the patients in the intervention group were also performed on the patients in the control group at the same hours. IV fluid therapy was not administered to both groups before surgical intervention.
  Interventions: Procedure: control group
- whey intake (Experimental): Since whey powder contains 73.45 grams of carbohydrate per 100 grams, whey was given to the patients in this study, unlike OCS (Oral Carbohydrate Solution), as it met the requirement in the ERAS protocol that at least 45 g of oral carbohydrate solution can be given two hours before surgery. It was prepared at the bedside by the first investigator for the patients in the oral whey intervention group by mixing 54 grams of 70% demineralized whey powder taken from the herbalist into 600 ml of drinking water six hours before the surgery, and the patients were given 400 ml six hours before the surgery and 200 ml two hours before the surgery. They were given ml and allowed to drink. Before the surgery, the patients' hunger, thirst, blood glucose and nausea and vomiting levels were evaluated.
  Interventions: Dietary Supplement: whey intake group

INTERVENTIONS:
Dietary Supplement: whey intake group — It was prepared at the bedside by the first investigator for the patients in the oral whey intervention group by mixing 54 grams of 70% demineralized whey powder taken from the herbalist into 600 ml of drinking water six hours before the surgery, and the patients were given 400 ml six hours before the surgery and 200 ml two hours before the surgery. They were given ml and allowed to drink.
  Arms: whey intake
Procedure: control group — The patients were left fasting after 00:00.
  Arms: control group

SUMMARY:
Whey Intake Blood Glucose, Fasting, Thirst, Nausea, Vomiting Elective Hip Fracture Surgery

DETAILED DESCRIPTION:
The prolonged fasting period before surgery causes symptoms such as anxiety, hypoglycemia, increase in gastric volume, decrease in pH value, development of insulin resistance, thirst, feeling of hunger, hypovolemia, dehydration, headache, etc. in patients. For these reasons,Guidelines for Preoperative Nutrition in Children and Adults prepared by the European Society of Anesthesiologists, it was stated that solid foods six hours before surgery and clear liquids two hours before surgery could be consumed.In the accelerated recovery protocol (Enhanced Recovery After Surgery- ERAS), the preoperative fasting period before anesthesia is stated as two hours for liquid foods and six hours for solid foods (high level of evidence, strong level of recommendation).

Carbohydrate drinks act as a main meal in patients, increasing satiety and reducing insulin resistance. Carbohydrate drinks also increase the feeling of thirst and help to improve thirst sensitization. Therefore, it is recommended that patients should drink them before surgery. Carbohydrate-rich liquids that can be drunk up to two hours before elective surgery reduce fasting, thirst and postoperative insulin resistance and make the person feel good (evidence level 1++, recommendation grade A).

Hip fracture is a problem that increases with advanced age. It seems likely that the encounter with this problem and its costs will increase in the world due to the prolongation of life expectancy. Furthermore, the increased risk of osteoporosis due to increased sedentary life and malnutrition contribute to the development of this problem.Surgery is required in the treatment of 98% of elderly patients with hip fractures. Besides, the presence of chronic diseases in most elderly patients increases the risk of mortality and morbidity. Therefore, the risk of perioperative complications in elderly patients with hip fractures is a serious clinical problem.

Whey is a translucent, greenish-yellow liquid protein source obtained from the precipitation of casein in cheese or casein production. Similar in composition to milk, whey contains about half of the milk dry matter, almost all of the milk sugar, about 1/5 of the proteins and most of the B vitamins. After technological developments, whey is no longer considered as a waste but is used in industry. Many clinical trials have shown that whey is effective in the treatment of cancer, AIDS, hepatitis B, heart diseases and osteoporosis. 6 Prolonged preoperative fasting in elderly patients causes metabolic changes, and postoperative nausea and vomiting cause changes in blood glucose and prolonged hospital stay. When the literature was reviewed, it was observed that the number of studies on whey in preoperative oral carbohydrate intake, which is included in ERAS protocols in orthopedic patients, is very limited and academic studies are needed. This study was conducted to determine the effect of whey, as a different liquid other than oral carbohydrate liquids, on patients hunger, thirst, blood sugar and nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older,
* Belonging to ASA II or III group,
* Having HA surgery for the first time, and
* Having the surgery performed under spinal anesthesia.

Exclusion Criteria:

* Diabetes Mellitus,
* Undergoing emergency surgery,
* Having gastrointestinal and endocrine problems,
* Using medications that may affect blood sugar,
* Patients with psychiatric/neurological disorders, patients who need any fluid or blood in the preoperative period, whey allergy, and patients who have intensive care in the postoperative period

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
blood glucose | 12 week
  The value was measured with 1ml of blood from the patient's fingertip.

SECONDARY OUTCOMES:
Fasting, Thirst | 12 week
  Hunger and thirst status was evaluated with VAS.VAS is a scale with different names at both ends on a 10 cm long vertical or horizontal line (0 = no hunger - no thirst, 10 = most severe hunger - thirst
Nausea and Vomiting | 12 week
  The Postoperative Nausea And Vomiting Impact Scale was used.A score of five or more from the scale indicates "clinically significant nausea and vomiting".

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Njoroge G, Kivuti-Bitok L, Kimani S. Preoperative Fasting among Adult Patients for Elective Surgery in a Kenyan Referral Hospital. Int Sch Res Notices. 2017 Apr 12;2017:2159606. doi: 10.1155/2017/2159606. eCollection 2017. PMID 28487877
- [Result] 3. Özyürek P. Hastanın sıvı yönetimi. Turkiye Klinikleri Journal of Surgical Nursing- Special Topics 2016:2(2);24- 32.
- [Result] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Result] 31. Ayoğlu, H, Uçan, B, Taşçılar, Ö, Atik, L, Kaptan Macit, Y, Turan Özkoçak, I(2009). Preoperatif oral karbonhidrat solüsyonu kullanılmasının hasta anksiyetesi ve konforu üzerine etkileri. TARD,37(6), 374-82.
- [Result] Noblett SE, Watson DS, Huong H, Davison B, Hainsworth PJ, Horgan AF. Pre-operative oral carbohydrate loading in colorectal surgery: a randomized controlled trial. Colorectal Dis. 2006 Sep;8(7):563-9. doi: 10.1111/j.1463-1318.2006.00965.x. PMID 16919107
- [Result] Deng Y, Fang Y, Li H, Chen J, An J, Qiao S, Wang C. A preoperative whey protein and glucose drink before hip fracture surgery in the aged improves symptomatic and metabolic recovery. Asia Pac J Clin Nutr. 2020;29(2):234-238. doi: 10.6133/apjcn.202007_29(2).0004. PMID 32674229
- [Result] 6. Güzeler N. Esmek E. Kalender M. Peyniraltı Suyu Ve Peyniraltı Suyunun İçecek Sektöründe Değerlendirilme Olanakları. Çukurova Tarım Ve Gıda Bilimleri Dergisi.2017:32(2); 27-36
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21712716/